CLINICAL TRIAL: NCT07105800
Title: A Pilot Study of Dance Intervention for Enhancing Executive Function and Physical Performance in Cognitively Impaired Older Adults
Brief Title: Dance Intervention to Improve Executive Function and Physical Performance in Older Adults With Cognitive Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMU-JIRBN202507032
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Older Adults; Cognitive Impairment, Mild
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music-based dance intervention group (Experimental): The intervention group participated in a structured, nine-week group-based dance program designed to stimulate both cognitive and motor functions. Each 40-minute session was held twice per week and featured music-based rhythmic movement combined with fixed choreography. The dance routines emphasized perceptual-motor training through mutual physical guidance, spatial coordination, and social interaction among participants. The intervention aimed to enhance executive function, balance, and lower limb mobility by incorporating dual-task elements that challenge memory, attention, and physical control in a dynamic, enjoyable setting.
  Interventions: Behavioral: Music-based dance
- Control group (Active Comparator): The control group participated in a structured, nine-week lower limb exercise program that included intermittent strength and balance training. Sessions were delivered twice weekly through standardized, non-musical instructional videos to ensure consistency and minimize cognitive stimulation.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Music-based dance — The dance routines emphasized perceptual-motor training through mutual physical guidance, spatial coordination, and social interaction among participants. The intervention aimed to enhance executive function, balance, and lower limb mobility by incorporating dual-task elements that challenge memory, attention, and physical control in a dynamic, enjoyable setting.
  Arms: Music-based dance intervention group
Behavioral: Control — The training content is delivered through standardized, non-musical instructional videos. Participants in the control group follow fixed video demonstrations to perform functional lower limb exercises. The movement components include independent lower limb strength training and balance training.
  Arms: Control group

SUMMARY:
This pilot study investigates the effects of a music-based dance intervention on executive function and physical performance in middle-aged and older adults with cognitive impairment. Dance, as a form of dual-task training, integrates music, rhythmic movement, and cognitive-motor coordination. When combined with group interaction and partner-guided physical cues, it has the potential to enhance both cognitive and motor functions simultaneously.

The intervention features a simple, structured dance sequence designed to stimulate rhythm, attention, and coordination through music-based movement. This study aims to evaluate the feasibility and preliminary efficacy of this approach in improving executive function and lower limb physical performance among individuals with cognitive impairment.

DETAILED DESCRIPTION:
Mild Cognitive Impairment (MCI) is an age-related condition that affects memory, judgment, and motor performance, often leading to reduced independence and quality of life. Recent studies have emphasized the interrelationship between cognitive and motor functions, particularly in individuals with neurodegenerative conditions. Interventions that incorporate dual-task training, such as dance, have shown promise in enhancing both domains by combining rhythmic movement, memory recall, physical coordination, and social interaction.

Dance-based interventions, especially those integrating music, external cues, and partner interaction, engage multiple brain regions including the frontal cortex, cerebellum, and hippocampus. These programs stimulate sensory-motor integration and executive control, potentially improving attention, gait, balance, and cognitive flexibility. Existing evidence supports that rhythm- and music-based movement, when combined with cognitive tasks, can enhance brain function, promote emotional regulation, and improve daily functioning in cognitively impaired populations.

This study aims to examine the effects of a structured, music-based dance intervention on executive function and physical performance in middle-aged and older adults with cognitive impairment. The program integrates fixed dance routines with perceptual-motor training and social interaction.

A total of 50 middle-aged and older adults receiving outpatient rehabilitation at a medical center in northern Taiwan were recruited and randomly assigned to either the music-based dance intervention group (n = 25) or the control group (n = 25). The intervention group participated in a nine-week group-based program involving rhythmic movement, mutual physical guidance, and social interaction. The control group completed a nine-week lower limb intermittent exercise program guided by non-musical instructional videos.

Assessments were conducted at three time points: pre-intervention, mid-intervention, and post-intervention. Evaluation tools included:Four-Square Step Test (FSST), Functional Reach Test (FRT), Timed Up and Go - Cognitive (TUG-Cognitive), Montreal Cognitive Assessment (MoCA), Stroop Color and Word Test (SCWT), Modified Borg Rating of Perceived Exertion (RPE), Course feedback questionnaire. Descriptive statistics were used to summarize participant demographics. Repeated measures analysis of variance (ANOVA) was used to examine within-group and between-group differences over time. Statistical analyses were performed using SPSS Statistics 26.0, with the significance level set at α < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjective Cognitive Decline (SCD) with a score ≥5 on the SCD-Q9 questionnaire, or Mild Behavioral Impairment (MBI) with a score ≥7 on the MBI-Checklist, with symptoms persisting for more than three months.
* Ability to follow instructions.
* Ability to stand unsupported or with assistive devices for at least 10 minutes.
* Ability to walk at least 10 meters, either unsupported or with assistive devices.

Exclusion Criteria:-Age below 55 years.

* Severe visual or hearing impairment.
* Score <16 on the Montreal Cognitive Assessment (MoCA).
* Emotional or anxiety symptoms caused by psychiatric medications that significantly impair the ability to perform study-related motor tasks.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | Baseline, mid-intervention (week 5), and one week post-intervention (week 10)
  The Montreal Cognitive Assessment (MoCA) is a widely used screening tool for detecting Mild Cognitive Impairment (MCI). It evaluates seven cognitive domains through 12 subtests, including: visuospatial and executive Function (e.g., cube copying and clock drawing), naming (e.g., visual confrontation naming), attention and Concentration (e.g., digit span, vigilance tasks), language (e.g., sentence repetition and verbal fluency), abstract Reasoning (e.g., similarity identification), memory (immediate and delayed recall), orientation (temporal and spatial). A total score of 26 or above is considered within the normal cognitive range. According to previous studies, a cut-off score of 24 offers optimal discrimination for MCI, with a reported sensitivity of 92% and specificity of 78%.

SECONDARY OUTCOMES:
Four-Square Step Test | Baseline, mid-intervention (week 5), and one week post-intervention (week 10)
  The FSST assesses motor-cognitive integration and fall risk. Participants are instructed to step rapidly and safely over four squares formed by crossed floor tape in a specified sequence. The test requires directional changes, weight shifting, and quick stepping, engaging both lower limb motor control and executive attention. FSST is widely used in populations with balance impairments, including older adults, individuals with stroke, Parkinson's disease, vestibular disorders, and limb amputations. Cut-off times indicating elevated fall risk vary by population: >15 sec in older adults and stroke patients, >9.68 sec in Parkinson's disease, >12 sec in vestibular disorders, and >24 sec in amputees. The FSST demonstrates excellent test-retest reliability (ICC = 0.98) and inter-rater reliability (ICC = 0.99)
Timed Up and Go - Cognitive | Baseline, mid-intervention (week 5), and one week post-intervention (week 10)
  This test evaluates dual-task performance by measuring the time needed to stand up from a chair, walk 3 meters, turn, return, and sit down, while performing a cognitive task (counting backward by threes from a random number). It reflects motor-cognitive integration, especially executive function and attention. Times >15 seconds suggest increased fall risk. One practice trial is provided for instruction comprehension. The test takes approximately 3 minutes and demonstrates excellent test-retest reliability (ICC = 0.96) and strong criterion validity (r = 0.86-0.92)
Functional Reach Test | Baseline, mid-intervention (week 5), and one week post-intervention (week 10)
  The FRT evaluates stability by measuring the maximal forward reach distance while standing with arms extended at 90 degrees and feet shoulder-width apart. The final reach distance is calculated by subtracting the starting fingertip position (third metacarpophalangeal joint) from the furthest reach. Three trials are averaged. Distances <15 cm indicate high fall risk. Normative values: 14-17 in (ages 20-40), 13-16 in (ages 41-69), and 10-13 in (ages 70-87). The FRT takes approximately 5 minutes to complete and demonstrates strong reliability (test-retest ICC = 0.90-0.95, inter-rater ICC = 0.89) and good face validity (r = 0.71)
Stroop Color and Word Test | Baseline, mid-intervention (week 5), and one week post-intervention (week 10)
  The SCWT measures selective attention, cognitive flexibility, and inhibitory control. It includes three parts: (1) reading color words, (2) naming colored squares, and (3) naming the ink color of incongruent color words (e.g., the word "red" printed in blue ink should be answered as "blue"). Each part is timed for 45 seconds, and performance is scored by the number of correct responses. The test demonstrates high internal consistency (ICC = 0.91), indicating strong reliability
Course Feedback Questionnaire | One week post-intervention (week 10)
  A custom three-item questionnaire developed to collect participant feedback on program experience and perceived benefits. Responses provide qualitative insight into engagement, satisfaction, and perceived change.

CONTACTS AND LOCATIONS:
Overall Officials: Fen-Ling Kuo, Principal Investigator — Department of Physical Medicine and Rehabilitation, Shuang Ho Hospital, Taipei Medical University
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Woods B, Rai HK, Elliott E, Aguirre E, Orrell M, Spector A. Cognitive stimulation to improve cognitive functioning in people with dementia. Cochrane Database Syst Rev. 2023 Jan 31;1(1):CD005562. doi: 10.1002/14651858.CD005562.pub3. PMID 39804128
- [Result] Wang RY, Huang YC, Zhou JH, Cheng SJ, Yang YR. Effects of Exergame-Based Dual-Task Training on Executive Function and Dual-Task Performance in Community-Dwelling Older People: A Randomized-Controlled Trial. Games Health J. 2021 Oct;10(5):347-354. doi: 10.1089/g4h.2021.0057. Epub 2021 Sep 1. PMID 34491113
- [Result] Tsai JC, Chen CW, Chu H, Yang HL, Chung MH, Liao YM, Chou KR. Comparing the Sensitivity, Specificity, and Predictive Values of the Montreal Cognitive Assessment and Mini-Mental State Examination When Screening People for Mild Cognitive Impairment and Dementia in Chinese Population. Arch Psychiatr Nurs. 2016 Aug;30(4):486-91. doi: 10.1016/j.apnu.2016.01.015. Epub 2016 Jan 21. PMID 27455923
- [Result] Sanprakhon P, Suriyawong W, Longphasuk N, Khatichop N, Arpaichiraratana C, Wongwiseskul S, Rattanaselanon P, Pipatpiboon N, Thaipisuttikul P. Effects of traditional Thai folk dance combined with cognitive stimulation program on behavior and cognition among older adults with cognitive decline: A randomized controlled trial. J Prev Alzheimers Dis. 2025 Apr;12(4):100066. doi: 10.1016/j.tjpad.2025.100066. Epub 2025 Jan 17. PMID 39824702
- [Result] Outermans JC, van Peppen RP, Wittink H, Takken T, Kwakkel G. Effects of a high-intensity task-oriented training on gait performance early after stroke: a pilot study. Clin Rehabil. 2010 Nov;24(11):979-87. doi: 10.1177/0269215509360647. Epub 2010 Aug 18. PMID 20719820
- [Result] McGirr A, Nathan S, Ghahremani M, Gill S, Smith EE, Ismail Z. Progression to Dementia or Reversion to Normal Cognition in Mild Cognitive Impairment as a Function of Late-Onset Neuropsychiatric Symptoms. Neurology. 2022 May 24;98(21):e2132-e2139. doi: 10.1212/WNL.0000000000200256. Epub 2022 Mar 29. PMID 35351783
- [Result] Lazarou I, Parastatidis T, Tsolaki A, Gkioka M, Karakostas A, Douka S, Tsolaki M. International Ballroom Dancing Against Neurodegeneration: A Randomized Controlled Trial in Greek Community-Dwelling Elders With Mild Cognitive impairment. Am J Alzheimers Dis Other Demen. 2017 Dec;32(8):489-499. doi: 10.1177/1533317517725813. Epub 2017 Aug 25. PMID 28840742
- [Result] Ilardi CR, Federico G, La Marra M, Amato R, Iavarone A, Soricelli A, Santangelo G, Chieffi S. Deficits in reaching movements under visual interference as a novel diagnostic marker for mild cognitive impairment. Sci Rep. 2025 Jan 14;15(1):1901. doi: 10.1038/s41598-025-85785-7. PMID 39805990
- [Result] Hao L, Jia J, Xing Y, Han Y. An application study-subjective cognitive decline Questionnaire9 in detecting mild cognitive impairment (MCI). Aging Ment Health. 2022 Oct;26(10):2014-2021. doi: 10.1080/13607863.2021.1980860. Epub 2021 Sep 29. PMID 34583593
- [Result] Chang CF, Yang RJ, Chang SF, Chou YH, Huang EW. The Effects of Quality of Life and Ability to Perform Activities of Daily Living on Mild Cognitive Impairment in Older People Living in Publicly Managed Congregate Housing. J Nurs Res. 2017 Jun;25(3):187-197. doi: 10.1097/JNR.0000000000000149. PMID 28481814
- [Result] Cao K, Bay AA, Hajjar I, Wharton W, Goldstein F, Qiu D, Prusin T, McKay JL, Perkins MM, Hackney ME. Rationale and Design of the PARTNER Trial: Partnered Rhythmic Rehabilitation for Enhanced Motor-Cognition in Prodromal Alzheimer's Disease. J Alzheimers Dis. 2023;91(3):1019-1033. doi: 10.3233/JAD-220783. PMID 36530084
- [Result] Bracco L, Pinto-Carral A, Hillaert L, Mourey F. Tango-therapy vs physical exercise in older people with dementia; a randomized controlled trial. BMC Geriatr. 2023 Oct 24;23(1):693. doi: 10.1186/s12877-023-04342-x. PMID 37875856
- [Result] Bisbe M, Fuente-Vidal A, Lopez E, Moreno M, Naya M, de Benetti C, Mila R, Bruna O, Boada M, Alegret M. Comparative Cognitive Effects of Choreographed Exercise and Multimodal Physical Therapy in Older Adults with Amnestic Mild Cognitive Impairment: Randomized Clinical Trial. J Alzheimers Dis. 2020;73(2):769-783. doi: 10.3233/JAD-190552. PMID 31868666